CLINICAL TRIAL: NCT02641288
Title: Intraperitoneal Ropivacaine Irrigation in Patients Undergoing Bariatric Surgery
Brief Title: Intraperitoneal Ropivacaine Irrigation in Bariatric Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Principal investigator, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HURJC15-77
Record Dates: First submitted 2015-12-18; First posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-12

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine irrigation (Experimental): Using a standard irrigation device, 300 mg total of ropivacaine in 200ml normal saline will be instilled into the abdomen after surgical dissection, just before abdominal wall closure. Under direct visualization, the solution is delivered over the oesophageal hiatus, over both anastomoses and in both subdiaphragmatic spaces.
  Interventions: Drug: Ropivacaine irrigation
- Normal saline irrigation (Placebo Comparator): Using a standard irrigation device, 200ml normal saline will be instilled into the abdomen after surgical dissection, just before abdominal wall closure. Under direct visualization, the solution is delivered over the oesophageal hiatus, over both anastomoses and in both subdiaphragmatic spaces.
  Interventions: Drug: Normal saline irrigation

INTERVENTIONS:
Drug: Ropivacaine irrigation — Using a standard irrigation device (no specific device is being used), 300 mg total of ropivacaine in 200ml normal saline will be instilled into the abdomen after surgical dissection, just before abdominal wall closure. Under direct visualization, the solution is delivered over the oesophageal hiatus, over both anastomoses and in both subdiaphragmatic spaces.
  Other Names: Intraperitoneal Ropivacaine irrigation
  Arms: Ropivacaine irrigation
Drug: Normal saline irrigation — Using a standard irrigation device (no specific device is being used), 200ml normal saline will be instilled into the abdomen after surgical dissection, just before abdominal wall closure.
  Other Names: Intraperitoneal Normal saline irrigation
  Arms: Normal saline irrigation

SUMMARY:
A prospective randomized clinical trial of all the patients undergoing laparoscopic sleeve gastrectomy (LSG) or laparoscopic Roux-en-Y gastric bypass (LRYGB) will be performed. Patients will be randomized in 2 groups: those patients undergoing intraperitoneal ropivacaine irrigation (Experimental Group - EG) and those undergoing intraperitoneal irrigation with normal saline (Control Group - CG).

DETAILED DESCRIPTION:
A prospective randomized clinical trial of all the patients undergoing laparoscopic sleeve gastrectomy (LSG) or laparoscopic Roux-en-Y gastric bypass (LRYGB) will be performed. Patients will be randomized in 2 groups: those patients undergoing intraperitoneal ropivacaine irrigation 300mg in 200 ml(Experimental Group - EG) and those undergoing intraperitoneal irrigation with normal saline 200ml (Control Group - CG).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >40 Kg/m2
* BMI > 35 Kg/m2 with the presence of comorbidities associated to obesity.

Exclusion Criteria:

* patients undergoing other bariatric techniques or revisional surgery
* allergy to local anesthetics
* severe underlying cardiovascular diseases
* chronic renal failure
* hepatic dysfunction
* previous foregut surgery
* patients with any contraindication for bariatric surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Pain | 24 hours postoperatively
  Postoperative pain will be evaluated by a blinded nurse 24 hours after surgery. Pain will be quantified using a visual analogic scale (VAS), ranging from 0(absence of pain) to 10 (unbearable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Gonzalez, MD, Study Director — Hospital General Elche

REFERENCES:
- [Derived] Ruiz-Tovar J, Gonzalez J, Garcia A, Cruz C, Rivas S, Jimenez M, Ferrigni C, Duran M. Intraperitoneal Ropivacaine Irrigation in Patients Undergoing Bariatric Surgery: a Prospective Randomized Clinical Trial. Obes Surg. 2016 Nov;26(11):2616-2621. doi: 10.1007/s11695-016-2142-z. PMID 27007272